CLINICAL TRIAL: NCT04413864
Title: Immunomodulatory Profile of Dexmedetomidine Sedation in Patients Recovering After ARDS Covid-19
Acronym: DEXDO-COVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP200413; 2020-A00799-30 (Other: ANSM)
Record Dates: First submitted 2020-04-21; First posted 2020-06-04 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-05

CONDITIONS: SARS-CoV 2
Keywords: SARS-CoV-2; Covid-19; Dexmedetomidine; Neuroinflammation
MeSH Terms: conditions — COVID-19; Neuroinflammatory Diseases

STUDY DESIGN:
Intervention Model Description: open-label monocentric cohort study, with intervention added
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SARS-CoV-2 (Covid-19 positive) (Other): Patients hospitalized in intensive care unit (ICU), infected with SARS-CoV-2
  Interventions: Other: Inflammatory cytokines and chemokines profiles of patients with dexmedetomidine administration

INTERVENTIONS:
Other: Inflammatory cytokines and chemokines profiles of patients with dexmedetomidine administration — Assigned Interventions:
  * Blood samples collection at inclusion (D0) and follow-up visits (D2, D7 and M6)
  * CAM-ICU scores during ICU hospitalisation, neurological questionnaires at M6 (GOAT, GOSE, MOCA, Barthel Index, PTSD, GDS, Rankin score, HADS)

SUMMARY:
Covid-19 infection is due to SARS-CoV-2 member of the Coronavirus family represented by SARS- and MERS-CoVwith neuronal tropism capacity for the brainstem and thalami. Dexmedetomidine has(i) central antihypertensive (ii) sedative and (iii) neuroprotective properties and is often used during patient recovering after mechanical ventilation withdrawal.

Dexmedetomidine administration could change the immunomodulatory profile of Covid-19 patients and reduce inflammatory response.CAM-ICU scores and Blood samples from Covid-19 ICU patients will be collected at 4 different timepoints (before Dexmedetomidine administration, at D2, D7 and M6) to analyse the inflammatory profile with different approaches:i) chromatin accessibility, ii) transcriptome analysis, iii) inflammatory cytokines and chemokines levels.

DETAILED DESCRIPTION:
Coronaviruses (CoV) cause enteric and respiratory diseases. Most human CoVs, such as hCoV - 229E, OC43, NL63 and HKU1, cause mild respiratory disease, but the global spread of two previously well-knownCoVs: Severe Acute Respiratory Syndrome (SARS-CoV) and Middle East respiratory syndrome (MERS-CoV) has proven the lethal potential of human CoV.

While MERS-CoV is still not eliminated from the world, another highly pathogenic CoV, currently named SARS- CoV-2, started in December 2019 in Wuhan, in China. This new CoV caused a Chinese outbreak of severe pneumonia (coronavirus 2019 [COVID - 19]), and quickly spread to other countries.

Genomic analyzes show that SARS-CoV-2 shares a highly homological sequence with other beta-coronavirus (βCoV) as MERS-CoV and SARS-CoV.

Some work published in the 2000s has shown the presence of SARS-CoV viruses in neurons. Similarly, some experimental work has demonstrate that the MERS-COV5 and SARS-CoV6 viruses detected in the intra-nasal airways have an affinity for several brain regions such as brainstem or thalami. MERS-Cov viral particles have been found in several organs, including brain after injection of an inoculum in mice.

Several studies indicate that the brain region involved in this context is the brainstem.

The path taken by the virus is not yet clear, but several arguments in the literature indicate the hematogenous or lymphatic pathway, in particular during the acute phase of the infection. In addition, a viral invasion of the peripheral nerves could occur, followed by a secondary cerebral invasion with synaptic transmission already shown for other viruses. Epidemiological data for SARS-CoV-2 (COVID-19 infection) showing median time between first symptoms and dyspnea of 5 days, and hospitalization of 7 days10. This delayed period seems sufficient to allow the virus to invade the central nervous system. A recent work shows that patients infected with COVID-19 have neurological symptoms (headache, nausea, vomiting).

Large doses of sedation could be required to control a phase of severe delirium found in Covid-19 positive patients during the recovering phase in ICU. This delirium could be explained by the manifestation of septic encephalopathy, or even direct spread of the virus in the central nervous system. Study of neuroinflammation biomarkers in bleed could understand the progression of the disease and propose therapeutic strategies according to the patient phenotype. In this context, the idea of finding a neuroprotective treatment to limit the toxic effect of this virus on the brain is promising.

Dexmedetomidine is a selective adrenergic receptor agonist with antihypertensive, hypnotic and analgesic properties. This molecule has an important capacity of diffusion in the central nervous system with a central action in the locus cœruleus involved in vigilance thus explaining its sedative action; it also acts on the posterior grey column also providing analgesia via hyperpolarization of nerve fibers type C. Its distribution and its elimination are done according to a bicompartmental model. It is strongly linked to plasma proteins (94%) and is metabolized by the liver by glucuronidation, with an elimination half-life of two hours, 90% eliminated by the kidney and 10% in the stool. Dexmedetomidine is a powerful sympatholytic and should never be administered as a bolus or as a loading dose, it should be administered as a continuous infusion at a start dose of 0.7 µg / kg / min and then adjusted to sedation scores between 0,4 and 1,1 µg/kg/h.

Dexmedetomidine has neuroprotective effects. In experimental models such as the intraperitoneal injection of LPS, spinal cord lesions and ischemia-reperfusion, dexmedetomidine lower the cerebral inflammation directly on the microglial phenotype. The molecular pathway involved is not clear yet, however several studies show an action of Dexmedetomidine on the MAP kinase pathway.

Dexmedetomidine could be a direct neuroprotective agent by decreasing the brain inflammation induced by Covid-19 infection. Adapted utilisation of Dexmedetomidine for each patient profile could facilitate recovery and shorten the stay of patients in intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years at time of inclusion
* Hospitalized in intensive care unit (ICU)
* Administration of dexmedetomidine scheduled for 7 days
* Intubated/ventilated patient infected with SARS-CoV-2 (Covid-19 positive patient)
* Patient affiliated to a social security system (French State medical aid excluded)
* Hemoglobin level ≥ 9 g /dL
* Patient or parent / close / trusted person having been informed about the study and having given informed consent (or inclusion procedure in an emergency situation)

Exclusion Criteria:

* Protected major (under safeguardship, curatorship or guardianship)
* Pregnancy or breastfeeding
* Contra-indication to dexmedetomidine administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04-24 (Actual); Primary Completion 2022-10-24 (Estimated); Study Completion 2022-10-24 (Estimated)

PRIMARY OUTCOMES:
Change of inflammatory cytokines concentration (mmol / L) in Covid19 + patients from Baseline at 6 months | Month6

SECONDARY OUTCOMES:
Change of interrelationship between inflammation (cytokines levels) and ICU delirium in Covid19 + patient from Baseline at 6 months | Month6
Modification in inflammatory genes expressed (expressed / non expressed) in PBMC between Baseline and M6 | Month6
Change in quantity of chromatine's openings (chromatin accessibility profiles) in ICU patient recovering from covid19 infection | Day2, Month6
Change in genes expression in Covid-19 patient with delirium in ICU between Day2 and Month6 | Day2, Month6

CONTACTS AND LOCATIONS:
Overall Officials: Vincent DEGOS, Pr, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Intensive Care Unit and Respiratory division ; Groupe hospitalier Pitie-Salpetriere and Universite Pierre et Marie Curie Paris 6, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided